CLINICAL TRIAL: NCT00937079
Title: The Physiology of Glucagon-like-peptide-1 Receptor Expression in Patients With Endogenous Hyperinsulinism - Correlation With Histopathology
Brief Title: Whole Body 111In-exendin-4 Imaging Study in Insulinoma Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Damian Wild, MD, University Hospital, Basel, Switzerland
Other Study IDs: OCS-01778-1
Record Dates: First submitted 2009-07-02; First posted 2009-07-10 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Hyperinsulinism; Hypoglycemia; Insulinoma
Keywords: Glucagon-like peptide-1 receptor targeting; Insulinoma imaging; Exendin-4; molecular imaging
MeSH Terms: conditions — Hyperinsulinism; Hypoglycemia; Insulinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor tissue
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: 111In-exendin-4 imaging — 90-100 megabecquerel (MBq) (30 microgram or less) 111In-exendin-4 IV once

SUMMARY:
The purpose of this study is to determine whether the investigators' new imaging modality (111In-exendin-4) has advantages in detecting insulinomas in comparison to conventional imaging.

DETAILED DESCRIPTION:
Insulinomas arise from pancreatic cells and are the most frequent hormone-active tumours of the pancreas. Insulinomas produce insulin and can become life threatening if they cannot be localised and removed surgically. Complete tumour resection cures most patients, hence surgery is the treatment of choice for begin and malignant insulinomas. The potential for surgical cure necessitates accurate tumour localisation before surgery because preoperative imaging facilitates the detection of small localised, multiple and metastatic insulinomas. However, the successful localisation of insulinomas is an challenging problem since approximately 30% of insulinomas cannot be visualised radiographically.

A novel nuclear medicine scanning method using radioactive exendin-4 (111In-exendin-4) has recently been developed for imaging of insulinomas. 111In-exendin-4 accumulates specifically in insulinoma cells via the glucagon-like peptide-1 (GLP-1) receptor. The accumulation of 111In-exendin-4 can be visualised by the use of a special camera (Single Photon Emission Computed Tomography (SPECT) camera) that detects radioactivity and lights up tumours as hot spots.

The decision to perform surgery is independent of this study. If surgery is performed a small sample of the tumor will be used for identifying the sites where 111In-exendin-4 binds to the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Biochemically proven endogenous hyperinsulinism confirmed by hypoglycaemia with neuroglycopenic symptoms, inadequately high serum insulin and C-peptide concentrations and negative sulfonylurea screening as well as low serum beta-hydroxybutyrate concentrations
* Able and willing to provide written informed consent

Exclusion Criteria:

* Renal insufficiency (creatinine > 140 micromol/l)
* Pregnancy or positive pregnancy test which will be performed in all patients without contraception and aged < 50 years
* Allergy to exendin-4 (Byetta®)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: residents of Switzerland
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Detection of insulinomas, cure rate | one year

CONTACTS AND LOCATIONS:
Overall Officials: Damian Wild, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Institute of Nuclear Medicine, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Result] Wild D, Macke H, Christ E, Gloor B, Reubi JC. Glucagon-like peptide 1-receptor scans to localize occult insulinomas. N Engl J Med. 2008 Aug 14;359(7):766-8. doi: 10.1056/NEJMc0802045. No abstract available. PMID 18703486
- [Result] Christ E, Wild D, Forrer F, Brandle M, Sahli R, Clerici T, Gloor B, Martius F, Maecke H, Reubi JC. Glucagon-like peptide-1 receptor imaging for localization of insulinomas. J Clin Endocrinol Metab. 2009 Nov;94(11):4398-405. doi: 10.1210/jc.2009-1082. Epub 2009 Oct 9. PMID 19820010